CLINICAL TRIAL: NCT03147040
Title: AssessinG Efficacy of Carboplatin and ATezOlizumab in Metastatic Lobular Breast Cancer: GELATO-trial
Brief Title: AssessinG Efficacy of Carboplatin and ATezOlizumab in Metastatic Lobular Breast Cancer
Acronym: GELATO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At interim analysis insufficient benefit was observed to continu the study
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M17GEL
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Lobular; Metastatic or incurable locally advanced cancer; Disease progression on endocrine therapy in advanced setting
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Carboplatin; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin/Atezolizumab (Experimental): Carboplatin AUC=1.5, weekly schedule, maximum 12 administrations Atezolizumab, 1200 mg flat dose, 3-weekly schedule, starting after two administrations of carboplatin
  Interventions: Drug: Carboplatin; Drug: Atezolizumab

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy treatment with carboplatin and atezolizumab
Drug: Atezolizumab — Chemotherapy treatment with carboplatin and atezolizumab

SUMMARY:
This is a single arm multicenter non-randomized phase II trial testing the efficacy of the combination of carboplatin plus atezolizumab in metastatic ILC

ELIGIBILITY:
Inclusion Criteria:

* Signed and written informed consent
* Age 18 year or older
* Metastatic or incurable locally advanced lobular breast cancer with confirmation of the lobular histology and E-cadherin loss on a biopsy of a metastatic lesion.
* Metastatic lesion accessible for histological biopsies
* Evidence of progression of disease
* A maximum of two lines of palliative chemotherapy
* WHO performance status of 0 or 1
* Evaluable disease or measurable according to RECIST 1.1

Exclusion Criteria:

* Leptomeningeal disease localization
* History of having received other anticancer therapies within 2 weeks of start of the study drug
* History of immunodeficiency, autoimmune disease, conditions requiring immunosuppression
* Prior treatment with immune checkpoint blockade
* Live vaccine within 2 weeks prior to start of study
* Active other cancer
* Active hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of patients free of progression at 6 months | At 6 months
  Progression as defined by RECST 1.1

SECONDARY OUTCOMES:
Number of patients free of progression at 6 months in the IR profile subgroup | At 6 months
  as defined by retrospective gene expression profiling
Number of patients free of progression at 6 months in the non- IR profile subgroup | At 6 months
  as defined by retrospective gene expression profiling
Number of patients free of progression at 12 months | At 12 months
  as defined by RECIST 1.1
Objective Response Rate | Assessed up to 60 months
  Number of patients with a partial or complete response
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Assessed up to one month after end of treatment
  Adverse events will be graded according to NCI Common Toxicity Criteria version 4.03
Overall Survival | Assessed up to 60 months
  time from start treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — NKI-AvL
Locations (4):
- Netherlands (4):
  - Antoni van Leeuwenhoek, Amsterdam
  - UMCG, Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center Cancer Institute, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided
to be decided

REFERENCES:
- [Derived] Voorwerk L, Isaeva OI, Horlings HM, Balduzzi S, Chelushkin M, Bakker NAM, Champanhet E, Garner H, Sikorska K, Loo CE, Kemper I, Mandjes IAM, de Maaker M, van Geel JJL, Boers J, de Boer M, Salgado R, van Dongen MGJ, Sonke GS, de Visser KE, Schumacher TN, Blank CU, Wessels LFA, Jager A, Tjan-Heijnen VCG, Schroder CP, Linn SC, Kok M. PD-L1 blockade in combination with carboplatin as immune induction in metastatic lobular breast cancer: the GELATO trial. Nat Cancer. 2023 Apr;4(4):535-549. doi: 10.1038/s43018-023-00542-x. Epub 2023 Apr 10. PMID 37038006